CLINICAL TRIAL: NCT05581940
Title: The Effect of Caudal Anesthesia Block on Perioperative Pain Control and Reduction of the Anesthetic Agent in Pediatric Infra-umbilical Surgery: A Prospective Randomized Trial Study
Brief Title: Pediatric Caudal Anesthesia Block. And Pain Control
Acronym: CEB
Status: Completed | Type: Observational
Sponsor: Salmaniya Medical Complex (Other Government)
Responsible Party: Principal Investigator, Zeana gawe, Specialist Of Anesthesia, Salmaniya Medical Complex
Other Study IDs: 123311219
Record Dates: First submitted 2022-07-31; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative; Adverse Reaction to Epidural Anesthesia; Anesthesia, Caudal
Keywords: caudal; Pain Management; Anesthesia; pediatric
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Analgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric caudal anesthesia block.: caudal epidural block is a neuraxial block to provide effective pain relief and analgesia in pediatrics undergoing infra-umbilical pediatric surgery this study aimed to compare the effectiveness of adding to general anesthesia in terms of Intra and post-op pain management. A prospective, randomized case-controlled.A total of 72 patients aged two months to six years with (ASA PS) I (ASA I) were recruited over a six-month period between December 2019 and May 2020. Patients were allocated into two groups A performed under general anesthesia with caudal block and group B performed under general anesthesia alone. Both groups were compared based on hemodynamic stability, analgesia need, pain score, and parental satisfaction. Postoperative pain was evaluated by the Pain Scale- Categorical and numerical variables of both groups were compared. Results:
  Interventions: Combination Product: Group A Caudal Epidural Anesthesia with bupivacaine 0.25% and group B with opioid intervenors

INTERVENTIONS:
Combination Product: Group A Caudal Epidural Anesthesia with bupivacaine 0.25% and group B with opioid intervenors — (CEB) in group A using drugs bupivacaine 0.25% commonly used in children including neonates in group A In infraumbilical operations, it is used as a supplement to GA and to control postoperative pain It is a safe, easy, and effective type of central neuraxial block.[ The patient will be intubated and the caudal block will be performed under GA after securing the airway. The patient's position will be turned onto the lateral decubitus then a landmark-based, blind technique will be used. In children, the success rate with the blind technique is above 96% but the occurrence of side effects is reported. Group B uses general anesthesia (GA) alone for intraoperative and perioperative pain control used the opioid intervious without caudal block .
  Other Names: Regional anesthesia intervention and pain control

SUMMARY:
Caudal epidural block CEB is the most commonly performed neuraxial block to provide effective pain relief and analgesia in patients undergoing infra-umbilical pediatric surgery. This study aimed to compare the effectiveness of adding CEB to general anesthesia in terms of intra- and post-operative pain management. Design: Double-unblinded.

Prospective. randomized. Study, Setting: salmanyia medical complex. intraoperative, postoperative recovery room Methods: A total of 72 patients American Society of Anesthesiology physical status classification ASA 1. Patients were equally allocated into two groups Group A and with CEB and Group B without CEB, aged two months to six years. respectively, over a study period of six months. Both groups were compared based on hemodynamic stability, level of sedation, analgesia need, pain score, and parental satisfaction. Postoperative pain was evaluated by four different pain scales.

DETAILED DESCRIPTION:
the data collection uses a combination of quantitative and qualitative data. Quantitative Data: These include numerical datasets, which can be analyzed with mathematical techniques and are collected based on scales such as numbers of patients with or without CEB, interval, ratio, and ordinal. Resultantly, then the data are surveys and questionnaires, observations of hemodynamics, and behaviors. and data pain scores are collected inside the recovery room and based on the Children's Hospital Eastern Ontario Pain Scale (CHEOPS), Faces Pain Scale-Revised (FPS-R), and Face, Legs, Activity, Cry CONSOL ability (FLACC) scales. That data was collected through four phases, pre-op Intra op and post-op 1 hour in PACU, and six hours post-op was observed by the nurses in the ward. the data is divided into primary and secondary. the primary data were directly collected from the parents and information on the medical history from the files in the hospital was recorded, and the secondary data was collected directly by the anesthesiologist inside the operation room Once the patient was shifted to the operating theatre, the patient's age, sex, weight, height, types of surgeries will be performed, and the type of GA induction and maintenance agents were recorded in the anesthesia charts then in the recovery room, patients, pain scores, and behaviors are monitored according to the regular in the organization, then in the ward are based on questionnaires, observations and comparing the statically significant value between the two groups. The raw data which was collected from case report forms were entered into a Microsoft Excel Spreadsheet initially. Then, the data have been transferred to and analyzed by IBM SPSS Statistics software version 21. The categorical and numerical variables of both groups were analyzed and compared. Data are expressed as n (%), mean ± standard deviation or median and interquartile range (IQR) according to distribution normality. Continuous variables were compared using the Mann-Whitney U test, and categorical variables were compared using Fisher's exact test or Pearson Chi-square test. The confidence interval was set at 95%.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between two months and six years
* who were undergoing infra-umbilical surgeries
* ASA PS I no any medical issues

Exclusion Criteria:

* CEB such as sacral anomaly
* bleeding diathesis, patients with neuromuscular disease,
* hemodynamically unstable were excluded from the study.
* Simple randomization was done to select patients who will receive CEB from the daily surgical list. This trial was not blinded.
* In terms of the sample size determination, for a study power of 80% and a probability of type I error of 5%, a total of 74 patients was required for the study.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: CONsolidated Standards of Reporting Trials (CONSORT) checklist was used for enrolment and allocation of patients. Children aged between two months and six years who were undergoing infra-umbilical surgeries with ASA PS I were randomly allocated to either group A (GA with CEB) or to group B (GA without CEB).,
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
demographic data in two groups recorded and compared intra operation room. | Demographic data of children in both groups. Recorded through study completion, an average of 1 year".
  the patient's in two groups .The demographic data for all patients as age\months, sex\female ,male, weight( kilogram ,Height\centimeter were recorded in the anesthesia chart.
hemodynamics changed in Bothe groups intra op and one hour and six hours post op | through study completion, an average of 1 year". Measures of change in bassline of hemodynamic stability in both groups A and B Period preop and interop and post operation the data are presented as mean ± standard deviation .
  the Baseline Systolic and diastolic Blood Pressure pre operation and intraoperation and 60 minuet post operation have been recorded in group A and group B..
pain scores and sedation degree of children through one and six hours post operation in both groups | through study completion, an average of 1 year Continuous variables were compared period one hour and 6 hours post op using Mann-Whitney U.df=degree of freedom,
  pain scores at the various time points, and postoperative analgesia Based on the Face, Legs, Activity, Cry, consolability (FLACC) scale is a measurement used to assess pain for children between the age of 2 month and 7 years or individuals that are unable to communicate their pain .the scale is scored range from 0 to 10 with 0 is presenting no paint the scale has five criteria witch are each assigned a score of 0,1 or ,2,

SECONDARY OUTCOMES:
Differences in CHEOPS Score (4-13) d\through one hour and six hours post operation. between group A and B | through study completion, an average of 1 year pain scale that is used to assist the pain in children in bout groups.
  All Children have been observed by nurses and anesthesiologists in post anesthesia care unit using the children s Hospital Estern Ontario Pain ScaleCHEOPS is a behaviors pain scale in young children for evaluating postoperative pain it used to monitor the effectiveness of interventions for reducing the pain and discomfort .CHEOPS pain score is sum points for the all 6 parameters cry. facial. touch. legs. child verbal. Torso. the score ranging from 4 to 13 where is considered above 5 presented of pain .and the score recorded at the 30 minutes .and 60 minutes add to 6 hours post operation. Using Mann-Whitney U test and categorical variables were compared using *Fisher's exact test or †Pearson Chi-square test. P value is considered statistically significant and, degree of freedom, confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Zeana Gawe, specialist, Principal Investigator — salmanyia medical complex
Locations (1):
- Salmanyia Medical Complex, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: No
the research data is intended for this research only and not to share in another research .and data were analyzed according to the protocol

REFERENCES:
- [Background] Suresh S, Long J, Birmingham PK, De Oliveira GS Jr. Are caudal blocks for pain control safe in children? an analysis of 18,650 caudal blocks from the Pediatric Regional Anesthesia Network (PRAN) database. Anesth Analg. 2015 Jan;120(1):151-156. doi: 10.1213/ANE.0000000000000446. PMID 25393589
- [Result] Banerjee A, Das B, Mukherjee D, Khanra M. A study of the effect of caudal epidural block on bispectral index targeted propofol requirement in children: A comparative study. J Indian Assoc Pediatr Surg. 2015 Apr-Jun;20(2):77-81. doi: 10.4103/0971-9261.151551. PMID 25829671
- [Result] Shamim F, Ullah H, Khan FA. Postoperative pain assessment using four behavioral scales in Pakistani children undergoing elective surgery. Saudi J Anaesth. 2015 Apr-Jun;9(2):174-8. doi: 10.4103/1658-354X.152874. PMID 25829906
- [Result] Senoglu N, Senoglu M, Oksuz H, Gumusalan Y, Yuksel KZ, Zencirci B, Ezberci M, Kizilkanat E. Landmarks of the sacral hiatus for caudal epidural block: an anatomical study. Br J Anaesth. 2005 Nov;95(5):692-5. doi: 10.1093/bja/aei236. Epub 2005 Sep 9. PMID 16155035
- [Result] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Result] Ozen V, Yigit D. A comparison of the postoperative analgesic effectiveness of low dose caudal epidural block and US-guided dorsal penile nerve block with in-plane technique in circumcision. J Pediatr Urol. 2020 Feb;16(1):99-106. doi: 10.1016/j.jpurol.2019.10.020. Epub 2019 Oct 30. PMID 31759904
- [Result] Nikooseresht M, Hashemi M, Mohajerani SA, Shahandeh F, Agah M. Ultrasound as a screening tool for performing caudal epidural injections. Iran J Radiol. 2014 May;11(2):e13262. doi: 10.5812/iranjradiol.13262. Epub 2014 May 15. PMID 25035698
- [Result] Kim YH, Park HJ, Cho S, Moon DE. Assessment of factors affecting the difficulty of caudal epidural injections in adults using ultrasound. Pain Res Manag. 2014 Sep-Oct;19(5):275-9. doi: 10.1155/2014/679128. Epub 2014 Aug 11. PMID 25111987
- [Result] Shin SK, Hong JY, Kim WO, Koo BN, Kim JE, Kil HK. Ultrasound evaluation of the sacral area and comparison of sacral interspinous and hiatal approach for caudal block in children. Anesthesiology. 2009 Nov;111(5):1135-40. doi: 10.1097/ALN.0b013e3181bc6dd4. PMID 19809281
- [Result] Ben-David B, Vaida S, Gaitini L. The influence of high spinal anesthesia on sensitivity to midazolam sedation. Anesth Analg. 1995 Sep;81(3):525-8. doi: 10.1097/00000539-199509000-00017. PMID 7653816
- [Result] Joo J, Kim J, Lee J. The prevalence of anatomical variations that can cause inadvertent dural puncture when performing caudal block in Koreans: a study using magnetic resonance imaging. Anaesthesia. 2010 Jan;65(1):23-6. doi: 10.1111/j.1365-2044.2009.06168.x. Epub 2009 Nov 17. PMID 19922508
- [Result] Manchikanti L, Cash KA, Pampati V, McManus CD, Damron KS. Evaluation of fluoroscopically guided caudal epidural injections. Pain Physician. 2004 Jan;7(1):81-92. PMID 16868617
- [Result] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329

DOCUMENTS (3):
  • Study Protocol (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT05581940/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT05581940/SAP_001.pdf
  • Informed Consent Form (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT05581940/ICF_002.pdf